CLINICAL TRIAL: NCT06208943
Title: Neural and Cognitive Consequences of COVID-19 Survival
Status: Recruiting | Type: Observational
Sponsor: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Judith Ford, Staff Neuroscientist/Clinician Investigator, San Francisco Veterans Affairs Medical Center
Other Study IDs: CX002322
Record Dates: First submitted 2024-01-11; First posted 2024-01-17 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: COVID Long-Haul; COVID-19; COVID-19 Pandemic; Brain Fog; Memory Deficits; Concentration Ability Impaired; Fatigue
Keywords: EEG; fMRI; MRI; functional MRI; brain fog; long COVID; fatigue; difficulty concentrating; memory difficulty
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19; Mental Fatigue; Memory Disorders; Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood draw
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NeuroCOVID Group: Individuals (ages 18-70 years) who endorse a reported change in concentration, memory, feelings anxiety or depression since initial COVID infection.
  Interventions: Other: cross-sectional MRI and EEG assessments (NO INTERVENTION)
- COVID Control Group: Individuals (ages 18-70 years) who do not feel any different since recovering from initial COVID infection.
  Interventions: Other: cross-sectional MRI and EEG assessments (NO INTERVENTION)

INTERVENTIONS:
Other: cross-sectional MRI and EEG assessments (NO INTERVENTION) — n/a there is no intervention in this observational study
  Other Names: cross-sectional MRI and EEG assessments

SUMMARY:
The novel coronavirus SARS-CoV-2 infection, COVID, continues to rage throughout the world with 115,000,000 confirmed cases and over 2,500,000 deaths (as of Mar 3, 2021). This translates to millions of people surviving COVID19 infection. While the lungs are ground zero, COVID tears through organ systems from brain to blood vessels. We are now beginning to see people recover but complain of ongoing problems, including lingering cognitive problems, depression, and anxiety. We have brought together 2 laboratories with complementary techniques including psychological testing and neuroimaging methods togethers with markers in the blood that may signal damage in the brain. A close look at these problems is timely and imperative if we are to understand the pathophysiology of 'COVID brain' and prepare for downstream problems.

DETAILED DESCRIPTION:
The SARS-CoV-2 pandemic has been going on for over a year worldwide, with 115,000,000 confirmed cases and over 2,500,000 deaths (as of Mar 3, 2021). We are seeing people recover from the initial COVID infection with complaints of ongoing problems. An increasing number of people are complaining of cognitive deficits and depression/anxiety.

Methodologically, we have brought together two laboratories studying neurocognitive impairment using an EEG, MRI, and behavioral approach as well as laboratory-based data. This study queries neuropsychological functions in individuals using a neuropsychological battery, EEG-based measures, functional MRI (connectivity) and structural MRI (gray and white matter volumes, myelin, micro-bleeds). In addition, we have preliminary data to show a continued increase in plasma cytokines in COVID survivors. Plasma isolated neuronal enriched extracellular vesicles (nEVs) showed an increase in amyloid beta, neurofilament light and pT181-Tau, all proteins associated with neurodegeneration.

The overall aim is to determine the extent of cognitive, clinical, and neurological damage in people recovered from COVID.

ELIGIBILITY:
Inclusion Criteria:

* Our studies require some in-person visits to our research lab, located at 42nd Ave and Clement St in San Francisco.
* Because this study includes an MRI, part of the screening process will be to ensure you don't have any metal in your body, you do not have head or neck tattoos, and you are comfortable inside the MRI scanner.
* 18-70 years with a confirmed COVID infection at least 3 months ago.
* Negative metal screen for MRI safety
* Normal (or corrected to normal) vision

Exclusion Criteria:

* Past or present neurological problems (including seizures and head trauma resulting in neurological or cognitive symptoms)
* Loss of consciousness (LOC) greater than 30 minutes or any LOC with neurologic symptoms
* Major medical conditions (e.g., seizures disorders, treatment with anticonvulsant medication, endocrine disorders, significant cardiac pathology)
* Substance dependence, within the past year, or failed urine toxicology on the day of neuroimaging sessions
* Known claustrophobia
* Current pregnancy
* IQ estimate < 70

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals 18-70 years old who were diagnosed with COVID-19 at least 3 months ago.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Change of Neuropsychological Test Performance | 1 month
  We will compare NP test performance in people with Covid-related worsening of attention, memory, anxiety, and/or depression to people who do not endorse worsening in those domains.
Number of Participants with EEG Latency & Amplitude | 1 month
  We will compare EEG-derived event related potential measures of neural speed in people with Covid-related worsening of attention, memory, anxiety, and/or depression to people who do not endorse worsening in those domains.
Number of Participants with MRI Functional Disconnectivity | 1 month
  We will compare thalamo-cortical connectivity in people with Covid-related worsening of attention, memory, anxiety, and/or depression to people who do not endorse worsening in those domains.
Number of Participants with Blood Biomarkers | 1 month
  We will correlate blood biomarkers of inflammation and NP test performance, thalamo-cortical connectivity, and measures of neural speed.

CONTACTS AND LOCATIONS:
Overall Officials: Judith M Ford, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco Heathcare System, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Not part of currently approved protocol or original agreement with sponsor.